CLINICAL TRIAL: NCT07032883
Title: Benson Relaxation Technique Effectiveness on Pain and Quality of Life Post Reconstructive Mammoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El-Monem Morad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005668
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benson relaxation technique and routine physiotherapy program group (Experimental): This group will receive Benson relaxation technique for duration up to 20 min twice daily in addition to medical therapy and a routine physical therapy program for 40 minutes, twice daily for 4 weeks.
  Interventions: Other: Benson relaxation technique; Other: Routine physiotherapy program; Drug: Medications
- routine physiotherapy program group (Active Comparator): This group will receive medical therapy and a routine physical therapy program for 40 minutes, twice daily for 4 weeks.
  Interventions: Other: Routine physiotherapy program; Drug: Medications

INTERVENTIONS:
Other: Benson relaxation technique — It will be performed every day, twice daily (in the morning and evening), for 4weeks, the Benson relaxation technique instruction included these steps.
  1. Sit in a comfortable position.
  2. Close their eyes.
  3. Relax all their muscles beginning from the soles of the feet, moving forward up, and relax all parts of their body.
  (4 ) Breath through their nose, pay attention to the sound of their breathing, and say the word ''one'' quietly to themselves when the breath is out.
  (5) Continue for 20 min. the patients were instructed to check the time by opening their eyes. However, using an alarm was prohibited. The training sessions were held during the patients hospitalization period after one week from surgery, the technique continued during the hospitalization and after discharge from the hospital.
  Arms: Benson relaxation technique and routine physiotherapy program group
Other: Routine physiotherapy program — The participants will receive routine physical therapy program (gentle stretching, manual therapy, mobility and strengthening exercises and posture training) for 40 minutes , for 4 weeks.
Drug: Medications — the participants will receive the following medications:
  1. Antibiotic: Ancef 1 g intravenous (IV) ( cefazolin) intravenous post-surgery every 8 hours for 24 hours. If allergic to ampicillin /cephalosporins clindamycin IV 600_900 mg every 8 hours for 24 hours. Then continue oral with keflex 1g tablets (cephalexin) twice daily for 7 days.
  2. Anti-inflammatory:
     Adolor ( ketorolac) 15_30 mg IV every 6 hours up to 5 days post-operation ( not exceed 120 mg/day) then followed by oral celecoxib 200 mg once or twice daily till pain subsides.
  3. paracetamol 500_1000 mg I.V every 6 hours for 5 days (Not exceed 4000 mg / day) Then followed by oral paracetamol tablets till pain subsides.
  4. Zurcal 40 mg IV (pantoprazol) then followed by oral zurcal tablets.

SUMMARY:
The purpose of this study is to evaluate effectiveness of benson relaxation technique on pain and quality of life post mammoplasty.

DETAILED DESCRIPTION:
Pain post reconstructive mammoplasty is common and has an impact on psychosocial aspects, anxiety, sleep disorders and activities of daily living(ADL),as a result patients suffer from impairment in quality of life.

To manage pain pharmaceutical and non-pharmaceutical interventions could be used.

Benson relaxation is a deep breathing relaxation therapy that has been developed by involving a person's belief factor. It works by shifting the focus of pain so that the body becomes relaxed, this can increase endogenous analgesics and be strengthened again by reciting spiritual sentences that provide calm.

Benson relaxation technique has a major effect on reducing anxiety, depression, and improving quality of life and psychological factors. Furthermore, this technique is easy to learn and no side effects have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Only female patients underwent reconstruction mammoplasty will participate in the study.
* Female patients who stopped chemotherapy at least one month before participation in the study.
* Female patients with chronic pain following cosmetic breast surgery.
* All patients who will accept to participate in the study after one week from operation.

Exclusion Criteria:

* Patients have irritable bowel syndrome.
* Patients have urinary incontinence.
* Chronic diseases like multiple sclerosis, polyneuropathy , diabetes and fibromyalgia.
* Patients have cognitive disorder.
* Patients with chronic and severe back pain.
* Sepsis with complications postoperative hemodynamics.
* Patients take anti-psychotic drugs.
* Patients take hypnotic drugs.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain severity | 4 weeks
  Visual analogue scale is a popularly used standardized scale for assessing pain intensity. It is 10 point horizontal line scale ranging from 0 to 10. The participants of both groups will be asked to mark the point representing their pain level before and after the intervention, with 0 meaning no pain and 10 meaning the worst pain.
Assessment of quality of life | 4 weeks
  The WHOQOL-BREF scale will be used to assess quality of life for all participants before and after the treatment program It is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. The highest possible score on the WHOQOL-BREF scale is 100. This score represents the best possible quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El Taher, Professor, Study Director — Ain Shams University; Haidy N Ashem, Professor, Study Chair — Cairo University
Locations (1):
- Mohamed Abd El-Monem Morad, Tanta, Egypt